CLINICAL TRIAL: NCT02976740
Title: A Prospective Multi-center Phase II Study: Assessment of the Safety and Abscopal Effects of SBRT Combination With rhGM-CSF and Thymosin Alpha 1 for Stage IV NSCLC Patients Who Failed in Second-line Chemotherapy
Brief Title: SBRT Combination With rhGM-CSF and Tα1 for Stage IV NSCLC Patients Who Failed in Second-line Chemotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KYZ2016-006
Record Dates: First submitted 2016-11-25; First posted 2016-11-29 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Lung Cancer Metastatic
Keywords: lung cancer; SBRT; rhGM-CSF; Thymosin Alpha 1
MeSH Terms: conditions — Lung Neoplasms | interventions — Adjuvants, Immunologic; Immunologic Factors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SBRT+GM-CSF+Tα1 (Experimental): Metastasis lesion will be treated with a SBRT of 50Gy/4-10F from day 1 to day 10 . Subcutaneous injection of Immunological Agent- human recombined granulocyte-macrophage colony stimulating factor (125ug/m² per day) will be executed from day 1 to day 14 in this cycle. Another metastasis lesion will be treated likewise concurrently with rhGM-CSF in a consecutive cycle. Subcutaneous injection of another Immunological Factors Thymosin Alpha 1(1.6mg Biw)will be executed from the fist WEEK to the 12th Weeks.
  Interventions: Radiation: SBRT; Drug: Immunological Agent; Drug: Immunological Factors

INTERVENTIONS:
Radiation: SBRT — Stereotactic body radiotherapy A type of radiation therapy to the Metastasis lesion
  Other Names: SABR
Drug: Immunological Agent — Subcutaneous injection of human recombined granulocyte-macrophage colony stimulating factor (125ug/m² per day) will be executed from day 1 to day 14 in this cycle. Another metastasis lesion will be treated likewise concurrently with rhGM-CSF in a consecutive cycle.
  Other Names: rh GM-CSF
Drug: Immunological Factors — Thymosin Alpha 1(1.6mg Biw)will be executed from the fist Week to the 12th Weeks.
  Other Names: Tα1

SUMMARY:
The purpose of this study is to determine whether stereotactic body radiotherapy (SBRT) combined with recombined human granulocyte-macrophage colony stimulating factor(rhGM-CSF) and Thymosin Alpha 1 is safe, effective in the treatment of stage IV NSCLC patients who failed in second-line chemotherapy.

DETAILED DESCRIPTION:
Metastasis lesion of stage IV NSCLC will be treated with a SBRT of 50Gy/4-10F from day 1 to day 14 in one cycle. Subcutaneous injection of human recombined granulocyte-macrophage colony stimulating factor (125ug/m² per day) will be executed from day 1 to day 14 in this cycle. Another metastasis lesion will be treated likewise concurrently with rhGM-CSF in a consecutive cycle.Thymosin Alpha 1(1.6mg Biw) will be Subcutaneous injection from the fist week to the 12th weeks, Efficacy evaluation, especially abscopal effect evaluation, will be conducted at the end of therapy and every month after that. Adverse events will be recorded according to NCI-CTC version 4.03.

ELIGIBILITY:
Inclusion Criteria:Inclusion Criteria:

1. Histologically proven non-small-cell lung cancer.
2. Stage IV according to UICC stage system(version 7,2009).
3. Progression after standard second-line chemotherapy.
4. At least Three evaluable lesions among which at least two must be suitable for SBRT.
5. ECOG performance status 0-2.
6. Expected lifespan ≥3 months.
7. Stable lab values:

   Hematological: Absolute neutrophil count (ANC) ≥1.5×109/L, Platelets ≥100×109/L, Hemoglobin ≥9 g/dL Renal: Creatinine OR Measured or calculated creatinine clearance (CrCl) (glomerular filtration rate [GFR] can also be used in place of creatinine or CrCl) ≤1.5× the upper limit of normal (ULN) OR ≥60 mL/min for patient with creatinine levels >1.5× institutional ULN Hepatic: Total bilirubin ≤1.5×ULN OR Direct bilirubin ≤ULN for patients with total bilirubin levels >1.5×ULN, Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5×ULN OR ≤5×ULN for patients with liver metastases ,globulin≥20 g/L, albumin≥30 g/L.
8. Female subjects must have a negative urine or serum pregnancy test within 72 hours prior to taking study drug if of childbearing potential.
9. Able to understand and give written informed consent and comply with study procedures.

Exclusion Criteria:

1. Any unstable systemic disease, including active infection, uncontrolled high blood pressure, unstable angina, newly observed angina pectoris within the past 3 months, congestive heart failure (New York heart association (NYHA) class II or higher), myocardial infarction onset six months before included into the group, and severe arrhythmia, liver, kidney, or metabolic disease in need of drug therapy, Including diabetes.
2. Any clinical evidence suggests moderately severe chronic obstructive pulmonary disease (COPD) - [With COPD history or related risk factors, FEV1 / FVC < 70%, FEV1 < 80% estimated value, with or without chronic cough, sputum, dyspnea symptoms), active interstitial lung disease - ILD (FEV1 / FVC < 70%, FEV1 < 80% estimated value, carbon monoxide diffusion capacity in lung - DLCO < 40%, and high resolution CT (HRCT) confirmed as the diffuse pulmonary interstitial lesions] and other active pulmonary disease.
3. Previously diagnosed with autoimmune diseases, including but not limited to systemic lupus erythematous, rheumatoid arthritis, systemic vasculitis, scleroderma, dermatomyositis, autoimmune hemolytic anemia and autoimmune liver disease, autoimmune thyroiditis.
4. Human immunodeficiency virus (HIV) infection.
5. Women in pregnancy or lactation .
6. Medicine abusers(including alcohol, drugs or other addictive drugs abusers).
7. Patients with mental illness, considered as "can't fully understand the issues of this research".
8. Cancer history within 5 years apart from NSCLC before enrollment.
9. Histologically confirmed small cell carcinoma or other non NSCLC compositions in the cancer tissue.
10. Cancer treatment within 4 weeks, including but not limited to palliative surgery ,radiotherapy, chemotherapy and target therapy.
11. Tumor related immunotherapy within 1 year, including but not limited to immune cell therapy, tumor vaccine therapy, immune check-point monoclonal antibody related treatment, and cytokines treatment except for GM-CSF.
12. Allergy of rhGM-CSF/Tα1 and its accessories.
13. Contraindications to GM-CSF/Tα1 treatment.
14. Patients with unilateral lung.

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2016-11; Primary Completion 2019-06 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
abscopal effect rate | at the time point of 4 weeks after completion of the combined treatment

SECONDARY OUTCOMES:
overall survival | 1 year after completion of the combined treatment
Incidence of Adverse events | 1 year after completion of the combined treatment
objective response rate | 4 weeks after completion of the combined treatment
Incidence of immune-related adverse events | 1 year after completion of the combined treatment

CONTACTS AND LOCATIONS:
Locations (1):
- First affiliated Hospital of Xiamen University, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Twyman-Saint Victor C, Rech AJ, Maity A, Rengan R, Pauken KE, Stelekati E, Benci JL, Xu B, Dada H, Odorizzi PM, Herati RS, Mansfield KD, Patsch D, Amaravadi RK, Schuchter LM, Ishwaran H, Mick R, Pryma DA, Xu X, Feldman MD, Gangadhar TC, Hahn SM, Wherry EJ, Vonderheide RH, Minn AJ. Radiation and dual checkpoint blockade activate non-redundant immune mechanisms in cancer. Nature. 2015 Apr 16;520(7547):373-7. doi: 10.1038/nature14292. Epub 2015 Mar 9. PMID 25754329
- [Background] Formenti SC, Demaria S. Systemic effects of local radiotherapy. Lancet Oncol. 2009 Jul;10(7):718-26. doi: 10.1016/S1470-2045(09)70082-8. PMID 19573801
- [Background] Mellman I, Coukos G, Dranoff G. Cancer immunotherapy comes of age. Nature. 2011 Dec 21;480(7378):480-9. doi: 10.1038/nature10673. PMID 22193102
- [Background] Zeng J, See AP, Phallen J, Jackson CM, Belcaid Z, Ruzevick J, Durham N, Meyer C, Harris TJ, Albesiano E, Pradilla G, Ford E, Wong J, Hammers HJ, Mathios D, Tyler B, Brem H, Tran PT, Pardoll D, Drake CG, Lim M. Anti-PD-1 blockade and stereotactic radiation produce long-term survival in mice with intracranial gliomas. Int J Radiat Oncol Biol Phys. 2013 Jun 1;86(2):343-9. doi: 10.1016/j.ijrobp.2012.12.025. Epub 2013 Feb 22. PMID 23462419
- [Background] Kalbasi A, June CH, Haas N, Vapiwala N. Radiation and immunotherapy: a synergistic combination. J Clin Invest. 2013 Jul;123(7):2756-63. doi: 10.1172/JCI69219. Epub 2013 Jul 1. PMID 23863633
- [Background] Suzuki Y, Mimura K, Yoshimoto Y, Watanabe M, Ohkubo Y, Izawa S, Murata K, Fujii H, Nakano T, Kono K. Immunogenic tumor cell death induced by chemoradiotherapy in patients with esophageal squamous cell carcinoma. Cancer Res. 2012 Aug 15;72(16):3967-76. doi: 10.1158/0008-5472.CAN-12-0851. Epub 2012 Jun 14. PMID 22700877
- [Background] Reits EA, Hodge JW, Herberts CA, Groothuis TA, Chakraborty M, Wansley EK, Camphausen K, Luiten RM, de Ru AH, Neijssen J, Griekspoor A, Mesman E, Verreck FA, Spits H, Schlom J, van Veelen P, Neefjes JJ. Radiation modulates the peptide repertoire, enhances MHC class I expression, and induces successful antitumor immunotherapy. J Exp Med. 2006 May 15;203(5):1259-71. doi: 10.1084/jem.20052494. Epub 2006 Apr 24. PMID 16636135
- [Background] Postow MA, Callahan MK, Barker CA, Yamada Y, Yuan J, Kitano S, Mu Z, Rasalan T, Adamow M, Ritter E, Sedrak C, Jungbluth AA, Chua R, Yang AS, Roman RA, Rosner S, Benson B, Allison JP, Lesokhin AM, Gnjatic S, Wolchok JD. Immunologic correlates of the abscopal effect in a patient with melanoma. N Engl J Med. 2012 Mar 8;366(10):925-31. doi: 10.1056/NEJMoa1112824. PMID 22397654
- [Result] Golden EB, Chhabra A, Chachoua A, Adams S, Donach M, Fenton-Kerimian M, Friedman K, Ponzo F, Babb JS, Goldberg J, Demaria S, Formenti SC. Local radiotherapy and granulocyte-macrophage colony-stimulating factor to generate abscopal responses in patients with metastatic solid tumours: a proof-of-principle trial. Lancet Oncol. 2015 Jul;16(7):795-803. doi: 10.1016/S1470-2045(15)00054-6. Epub 2015 Jun 18. PMID 26095785
- [Result] Golden EB, Demaria S, Schiff PB, Chachoua A, Formenti SC. An abscopal response to radiation and ipilimumab in a patient with metastatic non-small cell lung cancer. Cancer Immunol Res. 2013 Dec;1(6):365-72. doi: 10.1158/2326-6066.CIR-13-0115. PMID 24563870